CLINICAL TRIAL: NCT02633891
Title: Metabolic Syndrome and Fall Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F1651-W; 1IK2RX001651-01A2 (NIH)
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-03

CONDITIONS: Metabolic Syndrome; Autonomic Neuropathy
Keywords: neuropathies; metabolic diseases; nervous system diseases; peripheral nervous system diseases
MeSH Terms: conditions — Metabolic Syndrome; Metabolic Diseases; Nervous System Diseases; Peripheral Nervous System Diseases | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: parallel treatments
Who Masked: Outcomes Assessor
Masking Description: single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Balance exercise program (Experimental): Participants will attend weekly group training sessions and will keep an exercise log of home activity during a three month exercise program designed to improve balance. Balance exercises will be performed three times per week in a home-based training program.
  Interventions: Behavioral: Balance exercise
- standard care (Active Comparator): Participants will meet in person on a weekly basis for a general education class regarding health and fall prevention but will not participate in an exercise class.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Balance exercise — tailored balance exercise program
  Arms: Balance exercise program
Behavioral: Standard care — general health education and fall prevention classes
  Arms: standard care

SUMMARY:
Obesity and the metabolic syndrome (MetS) are rapidly growing problems. Individuals with the MetS are at risk for not only future chronic diseases, but they have a higher prevalence of neuropathy, including cardiac autonomic neuropathy, and have a higher incidence of falls. Currently there are no effective therapies to prevent or reverse the neuropathy seen in the MetS or to reduced the fall risk in this population. This research project will determine if a tailored balance exercise program will have functional benefits and result in a reduced fall risk in the growing population of patients with the MetS and neuropathy.

DETAILED DESCRIPTION:
Completed

55 participants with evidence of the MetS and autonomic neuropathy will be assessed for fall risk with the Four Square Step Test (FSST), which is a measure of dynamic standing balance. Additional endpoints include the dynamic gait index. Measures of height, weight, and waist circumference will be taken and an oral glucose tolerance test as well as lipids and blood pressure will also be measured. Autonomic function will be measured using cardiac autonomic testing, quantitative sudomotor axon reflex test and tilt table testing. Participants will be randomized into either a standard care group that will receive fall risk education or a targeted balance exercise intervention group. Both groups will meet once a week. The intervention group will receive a 12 week balance program with personalized incremental increases in the amount and difficulty of each maneuver.

ELIGIBILITY:
Inclusion Criteria:

* MetS at the time of screening based on the International Diabetes Federation definition
* No risk factors for other causes of neuropathy
* Autonomic neuropathy as defined by the Toronto Diabetic Neuropathy Expert Group 2010/11 consensus criteria
* Age 45-75 years inclusive at the time of screening
* Medically stable at the time of enrollment
* Able to participate in a standing balance exercise program without constant standby monitoring
* Women of childbearing potential must be using an acceptable method of contraception for the duration of their participation in the study
* Willing to accept assignment to either training group
* Willing and able to participate in the assigned intervention program

Exclusion Criteria:

* Pregnant women, prisoners, institutionalized subjects and other at risk subjects
* Etiology of neuropathy other than the MetS
* History of severe medical conditions likely to shorten lifespan or alter ability to participate in the trial
* Severe autonomic neuropathy that restricts daily function and the ability to participate in study interventions
* An inability to understand or cooperate with the procedures of the trial or refusal to sign the informed consent

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay A Zilliox, MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Balance Exercise Program | Standard Care
Started | 7 | 5
Completed | 5 | 4
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Balance Exercise Program | Standard Care | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Continuous [Mean (Full Range); unit: years] | 66 [53 to 74] | 66 [59 to 75] | 66 [53 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Full Range); unit: kg/m^2] | 35.64 [26.5 to 49.2] | 38.16 [29.9 to 47.4] | 36.69 [26.5 to 49.2]
Fasting glucose [Mean (Full Range); unit: mg/dL] | 133.86 [97 to 203] | 108.4 [91 to 130] | 123.25 [91 to 203]
Four square step test [Mean (Full Range); unit: seconds] | 14.49 [8.62 to 31.56] | 13.01 [8.15 to 22.6] | 13.91 [8.15 to 31.56]
Dynamic Gait Index (DGI) [Mean (Full Range); unit: score on a scale] — The short form DGI is scored 0-12, with higher number indicating better performance. It is used for the clinical assessment of walking function. Each of four items (horizontal head turns, vertical head turns, gait on level surfaces, and changes in gait speed) are scored on an ordinal scale from 0-3 with higher numbers indicating better performance.
  score on a scale | 7 [3 to 9] | 9 [5 to 12] | 7.73 [3 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Four Square Step Test (FSST)
Description: A measure of proactive dynamic standing balance. A participant steps over four canes that are laid on the ground at 90 degree angles to each other. The participants stands in one of the squares formed by the canes and they are instructed to step as quickly as possible into each square in a specified sequence.
Time Frame: 12 weeks
Population: In the balance exercise program 2 participants were lost to follow up and 2 participants did not complete the 12-week mobility testing, which included the FSST.
  In the standard care group 1 participant was lost to follow up.
Measure: Mean (Full Range); unit: seconds
Arm/Group | Balance Exercise Program | Standard Care
Number analyzed (Participants) | 3 | 4
seconds | 11.04 [9.9 to 12.93] | 14.29 [9.28 to 25.47]

2. Secondary Outcome: Dynamic Gait Index (DGI)
Description: An instrumented DGI will be performed on an instrumented gait mat. The DGI is a measure of functional balance during walking and it assesses an individual's ability to modify balance while walking in the presence of external demands (walking while changing speeds, head turns, stepping over and around obstacles, pivoting, and stair climbing).
  The short form DGI is scored 0-12, with higher number indicating better performance.
Time Frame: 12 weeks
Population: In the balance exercise program 2 participants were lost to follow up and 2 participants did not complete the 12-week mobility testing, which included the DGI.
  In the standard care group 1 participant was lost to follow up.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Balance Exercise Program | Standard Care
Number analyzed (Participants) | 3 | 4
score on a scale | 9.33 [8 to 10] | 7.5 [3 to 11]

ADVERSE EVENTS:
Time Frame: 3 years
Description: only deaths and serious adverse events were assessed. Other (not including serious) adverse events were not monitored/assessed.
Arm/Group | Balance Exercise Program | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-05-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT02633891/Prot_SAP_000.pdf
  • Informed Consent Form (2016-03-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT02633891/ICF_001.pdf